CLINICAL TRIAL: NCT04131907
Title: A Prospective, Multicenter, Double Blind, Randomized, Clinical Study to Evaluate the Safety and Efficacy of the Optilume™ BPH Catheter System in Men With Symptomatic BPH
Brief Title: Optilume™ BPH Catheter System in Men With Symptomatic BPH
Acronym: PINNACLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PR1087
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH, Drug Coated Balloon, DCB, prostate, LUTS, Optilume
MeSH Terms: conditions — Prostatic Hyperplasia; Color Vision Defects

STUDY DESIGN:
Intervention Model Description: Randomized study with a non-randomized, Pharmacokinetics arm. Subjects randomized to the Control arm are allowed to crossover to the Test arm if they meet the eligibility criteria after completing the 3-Month Follow-up Visit and prior to the close of the 12-Month visit window.
  Up to 625 subjects will be enrolled (i.e. consented) in the study in order to identify 162 eligible subjects (147 randomized subjects and 15 Pharmacokinetic subjects)
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects in the Randomization arm of the study are randomized in a 2:1 allocation of Test to Control. The treating physician is unblinded to the treatment assignment. A blinded person at the study site conducts all study follow-up visits through the 12-Month follow-up visit (or until the subject is unblinded). The subject may be unblinded prior to the 12-Month visit if it is medically necessary, which includes the subject seeking alternative BPH therapy due to continued or recurrent BPH symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Optilume™ BPH Catheter System (Experimental): The Optilume™ BPH, Prostatic Dilation DCB Catheter is a dilation catheter used to exert radial force to dilate the prostatic urethra resulting in a commissurotomy. The distal end of the catheter has a semi-compliant inflatable double lobe balloon that is coated with a proprietary coating containing the active pharmaceutical paclitaxel.
  Interventions: Device: Optilume BPH Catheter System
- Sham Device (Sham Comparator): The Sham Device is a 21 Fr Optilume BPH, Prostatic Pre-dilation Catheter within the sheath.
  Interventions: Device: Optilume Sham Device
- Pharmacokinetics Optilume Arm (Experimental): A single arm of 15 non-randomized subjects will be treated in the pharmacokinetics (PK) arm. These subjects will be treated with the Optilume BPH Catheter System
  Interventions: Device: Optilume BPH Catheter System

INTERVENTIONS:
Device: Optilume BPH Catheter System — The Optilume™ BPH, Prostatic Dilation DCB Catheter is a dilation catheter used to exert radial force to dilate the prostatic urethra resulting in a commissurotomy. The distal end of the catheter has a semi-compliant inflatable double lobe balloon that is coated with a proprietary coating containing the active pharmaceutical paclitaxel.
  Arms: Optilume™ BPH Catheter System; Pharmacokinetics Optilume Arm
Device: Optilume Sham Device — 21 Fr sheathed Optilume™ BPH Prostatic Pre-dilation Catheter (modified to prevent inflation)
  Arms: Sham Device

SUMMARY:
PINNACLE is a prospective, multi-center, randomized control clinical trial to establish the safety and efficacy of the Optilume™ BPH Catheter System in the treatment of benign prostatic hyperplasia (BPH)

DETAILED DESCRIPTION:
This is a prospective, multi-center, double blind, randomized controlled clinical trial in a 2:1 allocation of Test versus sham Control. In addition, a single arm of 15 non-randomized subjects will be added to study the Pharmacokinetics of the drug. The objectives of the study are to assess the efficacy of Optilume BPH Catheter System to alleviate LUTS believed to be secondary to BPH (LUTS/BPH) and to evaluate the safety of Optilume BPH Catheter System in the treatment of LUTS/BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject 50-80 years of age who has symptomatic BPH
2. International Prostate Symptom Score (IPSS) ≥ 13
3. Peak urinary flow rate (Qmax) ≥ 5 ml/sec and ≤ 12 ml/sec (with minimum voided volume of ≥ 150 ml)
4. Prostate volume 20 to 80 gm as determined by transrectal ultrasound (TRUS)
5. Prostatic urethral length ≥ 32 mm and ≤ 55 mm as determined by TRUS
6. History of inadequate response, contraindication, or refusal of BPH medical therapy
7. Able to complete the study protocol in the opinion of the investigator

Exclusion Criteria:

1. Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with all the follow-up requirements
2. Unwilling to abstain or use protected sex for the first 30 days post treatment
3. Unwilling to abstain from sexual intercourse or use a highly effective contraceptive for at least 6 months post-procedure
4. Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate
5. Any prior minimally invasive intervention (e.g. TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
6. Prostate specific antigen (PSA) ≥ 10 ng/ml unless prostate cancer is ruled out by biopsy
7. Confirmed or suspected malignancy of prostate or bladder
8. Active or history of epididymitis within the past 3 months
9. Previous pelvic irradiation or pelvic trauma surgery
10. Active urinary tract infection (UTI) confirmed by culture
11. Bacterial prostatitis within the last 12 months
12. Non-bacterial prostatitis within the last 5 years
13. Visible or invisible hematuria (> 4 Red Blood Cells (RBCs) per high power field) on 2 separate urine specimens within the last 3 months without a know contributing factor
14. Neurogenic bladder or sphincter abnormalities or neurological disorders that might affect bladder or sphincter function
15. History of urinary incontinence
16. Previous or current diagnosis of urethral strictures, bladder neck contracture or detrusor muscle spasms
17. Previous rectal surgery, other than hemorrhoidectomy
18. Use of antihistamines, anticonvulsants or antispasmodics within 1 week prior to baseline assessment unless there is documented evidence of stable dosing for at least 6 months
19. Use of antidepressants with adrenergic effects (i.e. duloxetine, imipramine and amitriptyline), long-acting anticholinergics (LAAC) for chronic obstructive pulmonary disease (COPD), or androgens within 2 weeks prior to baseline assessment unless there is documented evidence of stable dosing for at least 3 months prior to baseline assessment
20. Use of Luteinizing Hormone-Releasing Hormone (LHRH) analogs within 12 months prior to baseline assessment
21. Use of Type II 5-alpha reductase inhibitor [e.g. finasteride (Proscar, Propecia)] within 3 months of baseline assessment
22. Use of 5-alpha reductase inhibitor [e.g. dutasteride (Avodart)] within 6 months of baseline assessment
23. Use of estrogen or drugs producing androgen suppression unless there is documented evidence of stable dosing for at least 3 months prior to baseline assessment
24. Use of alpha blockers or daily dose PDE5 inhibitor (e.g. Cialis) within 2 weeks of baseline assessment
25. Use of warfarin or novel oral anti-coagulants [e.g., apixaban (Eliquis), fondaparinux (Arixtra), rivaroxaban (Xarelto) or edoxaban (Savaysa)], unless the medication is safely discontinued prior to the procedure and is not planned to be restarted for at least 5 days post-procedure
26. Use of anti-platelet medications (e.g., clopidogrel, aspirin) within 10 days prior to the procedure or planned use within 5 days post-procedure
27. History of hypersensitivity reactions to paclitaxel, on medication that may have negative interaction with paclitaxel, presence of solid tumor with a baseline neutrophil count of <1500 cells/mm3 or AIDS-related Kaposi's sarcoma with baseline neutrophil count of <1000 cells/mm3
28. Incidence of spontaneous urinary retention within 6 months prior to baseline assessment
29. Current post-void residual volume > 300 ml or catheter dependent bladder drainage
30. Known poor detrusor muscle function (e.g. Qmax < 5 ml/sec)
31. Current bladder or prostatic urethral stones
32. Biopsy of prostate within 40 days prior to procedure
33. History of cancer in non-genitourinary system which is not considered in complete remission (except basal cell or squamous cell carcinoma of the skin). A potential participant is considered in complete remission if there has been no evidence of cancer within five years
34. Current uncontrolled diabetes (i.e. hemoglobin A1c ≥ 8%)
35. History of clinically significant comorbidities or presence of unstable conditions [e.g. cardiovascular, lung, renal (serum creatinine > 2.0 mg/dl), hepatic, bleeding disorders or metabolic impairment] that may confound the results of the study or have a risk to subject per investigator's opinion
36. Any cognitive disorder that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affects the ability to complete the study quality of life questionnaires
37. Life expectancy < 10 years
38. Anatomy (e.g. presence of false passage or size of meatus) is not suitable for treatment in this study
39. Significant median lobe component [e.g. intravesical prostatic protrusion (IPP) > 1 cm]
40. Device that corresponds with the subject's prostate size is not available
41. Currently enrolled in or plan to enroll in another investigational clinical study for any disease except for observational only study
42. In the opinion of the investigator, it is not in the subject's best interest to participate in the study

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Kaplan, MD, Principal Investigator — Mount Sinai Health System
Locations (21):
- United States (19):
  - Arkansas Urology, Little Rock, Arkansas
  - Colorado Clinical Research, Golden, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - Florida Urology Partners, Tampa, Florida
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Sheldon Freedman MD, Ltd, Las Vegas, Nevada
  - New Jersey Urology, Englewood, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice, PLLC, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Associated Urologists of NC, Raleigh, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Austin, PLLC, Austin, Texas
  - North Austin Urology, Austin, Texas
  - Rio Grande Urology, El Paso, Texas
  - Clear Lake Specialties, Webster, Texas
- Canada (2):
  - University Urology Associates, Toronto, Ontario
  - University of Montreal Hospital Center (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaplan SA, Moss JL, Freedman SJ. Two-year long-term follow-up of treatment with the Optilume BPH catheter system in a randomized controlled trial for benign prostatic hyperplasia (The PINNACLE Study). Prostate Cancer Prostatic Dis. 2024 Sep;27(3):531-536. doi: 10.1038/s41391-024-00833-z. Epub 2024 Apr 29. PMID 38684918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 162 subjects will be randomized and/or treated in the study at up to 30 clinical sites in the United States and Canada. Up to 625 subjects will be enrolled (i.e. consented) in the study in order to identify 162 eligible subjects to be randomized and/or treated. All subjects treated with the Optilume BPH Catheter System will be followed annually through 5 years. Study duration is approximately 8 years.
Pre-assignment Details: Any required procedures performed before obtaining informed consent as part of the standard of care may be used in lieu of the study tests. Subjects who require a washout period should have these evaluations, with the exception of informed consent, conducted following completion of the washout period. Subjects who cannot tolerate a drug washout or are considered high risk from the drug washout should be excluded from the study.
Groups:
- TEST ARM - Optilume™ BPH Catheter Treatment in Men With Symptomatic BPH System: Subjects randomized to the Test arm were treated with the Optilume™ BPH Catheter System.
  Subjects were evaluated at baseline, immediately post-procedure, at Foley removal, 14 days, 30 days, 3 months, 6 months, 12 months and annually through 5 years post-procedure.
  Randomized subjects were blinded to the treatment assignment through the 12-month Follow-up Visit.
- CONTROL ARM - Sham Treatment in Men With Symptomatic BPH.: Subjects randomized to the Control arm received a sham procedure. A cystoscopy was performed followed by insertion of the sham device (21 Fr Optilume BPH, Prostatic Pre-dilation Catheter with a modified catheter hub to prevent inflation of the balloon) within the sheath.
  Subjects were evaluated at baseline, immediately post-procedure, at Foley removal, 14 days, 30 days, 3 months, 6 months and 12 months.
  Randomized subjects were blinded to the treatment assignment through the 12-month Follow-up Visit.
  Subjects randomized to the Control arm were allowed to crossover to the Test arm (treated with Optilume BPH) if they met the eligibility criteria after completing the 3-Month Follow-up Visit and prior to the close of the 12-Month visit window. Data for these subjects is reported seperately as the Crossover Cohort.
- Pharmacokinetic (PK) Arm: Subjects in the Pharmacokinetic (PK) arm of the study were not randomized and were treated with the Optilume BPH Catheter System.
  Small amounts of blood, urine and semen were collected for pharmacokinetic testing and sperm quality testing. Subjects are followed through 5-years post-procedure.
  A total of 15 subjects were included in the PK arm, with one of those subjects also being included in the Crossover cohort. For this summary of the study results, 14 subjects will be indicated as participating in the PK arm to prevent the PK Crossover subject from being counted twice in the numbers.
  A central core laboratory was utilized for analysis of the PK samples.
Period: Overall Study
Arm/Group | TEST ARM - Optilume™ BPH Catheter Treatment in Men With Symptomatic BPH System | CONTROL ARM - Sham Treatment in Men With Symptomatic BPH. | Pharmacokinetic (PK) Arm
Started | 100 (Subjects randomized to the Test arm will be treated with the Urotronic Optilume BPH Catheter System. For the Primary Endpoint, the analysis population will be intent to treat (ITT). Data from subjects randomized to this arm will be used in the analyses.) | 48 (Subjects randomized to the Control arm will receive a sham procedure. A cystoscopy will be performed followed by insertion of the 21 Fr Optilume BPH, Prostatic Pre-dilation Catheter within the sheath. The catheter hub of the sham device will be modified to prevent inflation of the balloon.) | 14 (A single arm of 14 non-randomized subjects will be treated in the pharmacokinetics (PK) arm. These subjects will be treated with the Optilume BPH Catheter System)
Crossover Cohort | 0 | 25 | 0
Completed | 90 | 26 | 12
Not Completed | 10 | 22 | 2
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 4 | 22 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Treatment failure | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pharmacokinetic (PK) Arm: A single arm of 14 non-randomized subjects will be treated in the pharmacokinetics (PK) arm.
  The Optilume™ BPH, Prostatic Dilation DCB Catheter is a dilation catheter used to exert radial force to dilate the prostatic urethra resulting in a commissurotomy.
- Total: Total of all reporting groups
Arm/Group | Optilume™ BPH Catheter System | Sham Device | Pharmacokinetic (PK) Arm | Total
Number analyzed (Participants) | 100 | 48 | 14 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: PK Arm added to Measure Analysis Population
  Years | 64.5 (6.4) | 65.5 (5.6) | 65.6 (7.4) | 64.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Endpoints will be analyzed using the Intent To Treat (ITT) population
  Participants
    number analyzed (Participants) | 98 | 48 | 14 | 160
    Female | 0 | 0 | 0 | 0
    Male | 98 | 48 | 14 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 3 | 0 | 16
  Not Hispanic or Latino | 87 | 45 | 14 | 146
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographics for PK Arm
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 2 | 0 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 5 | 1 | 9
    White | 94 | 43 | 12 | 149
    More than one race | 1 | 0 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 94 | 46 | 14 | 154
  Canada | 6 | 2 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With >30% Improvement in the International Prostate Symptom Score (IPSS)
Description: The primary efficacy endpoint was the improvement in International Prostate Symptom Score (IPSS) at 12 months in the Optilume BPH arm compared to the improvement in IPSS at 3 months in the Sham arm with a super-superiority margin on 25%.
  The IPSS contains the well-validated, highly reliable and responsive American Urological Association symptom score (AUASS) assessment to identify the severity of BPH symptoms. The first seven questions in the IPSS address frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying, and urgency, and scored on a 6-point scale (0 to 5). The IPSS can be interpreted as follows: 0-7 mildly symptomatic, 8-19 moderately symptomatic, and 20-35 severely symptomatic.
  The IPSS also includes an eighth question that is designed to assess the degree of "bother" associated with the subject's urinary symptoms. Answers range from "delighted" to "terrible" (0-6). This question is not included in the calculation of the main IPSS score.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume™ BPH Catheter System | Sham Device
Number analyzed (Participants) | 100 | 48
Participants | 89 | 26

2. Primary Outcome: Number of Participants With Major Device Related Serious Complications
Description: Rate of major device-related serious complications. A major device-related serious complication is defined as any of the following events through 12 months:
  * Device-related rectal fistula or GI fistula
  * Device-related formation of fistula between the rectum and urethra
  * Device-related new onset severe urinary retention lasting > 14 consecutive days post-healing
  * Device-related unresolved new onset stress urinary incontinence by 90 days
  * Device-related bleeding requiring transfusion
  * Device-related urethra or prostatic capsule rupture requiring surgical intervention
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume™ BPH Catheter System | Sham Device
Number analyzed (Participants) | 100 | 48
Participants | 89 | 26

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Optilume™ BPH Catheter Treatment in Men With Symptomatic BPH System: Subjects were randomized to treatment with the Optilume™ BPH Catheter System prior to study procedure.
- Sham BPH Catheter Treatment in Men With Symptomatic BPH.: Subjects randomized are blinded to the treatment assignment through the 12-month Follow-up Visit.
- Crossover Cohort: Subjects randomized to Sham who had ongoing or recurrent LUTS elected to receive the Optilume BPH Catheter System. Crossover to receive Optilume BPH was allowed before the close of the 12-month follow up period from randomization.
- Pharmacokinetic(PK): Subjects enrolled in the Pharmacokinetics arm of the study were be treated with the Optilume BPH Catheter System.
Arm/Group | Optilume™ BPH Catheter Treatment in Men With Symptomatic BPH System | Sham BPH Catheter Treatment in Men With Symptomatic BPH. | Crossover Cohort | Pharmacokinetic(PK)
All-Cause Mortality (participants affected / at risk) | 1/98 | 0/48 | 0/25 | 0/14
Serious Adverse Events (participants affected / at risk) | 14/98 | 3/48 | 0/25 | 0/14
Other Adverse Events (participants affected / at risk) | 81/98 | 14/48 | 15/25 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optilume™ BPH Catheter Treatment in Men With Symptomatic BPH System (N=98) | Sham BPH Catheter Treatment in Men With Symptomatic BPH. (N=48) | Crossover Cohort (N=25) | Pharmacokinetic(PK) (N=14)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA | NA
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | NA | NA
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | NA | NA
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | NA | NA
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Chest Pain (non cardiac (General disorders) | 1 (1) | 0 (0) | NA | NA
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA | NA
Cervical Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA
Suicidal Depression (Psychiatric disorders) | 1 (1) | 0 (0) | NA | NA
Bladder Perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | NA | NA
Post Procedural Hematuria (Renal and urinary disorders) | 4 (4) | 0 (0) | NA | NA
Urethral False Passage (Renal and urinary disorders) | 1 (1) | 0 (0) | NA | NA
Atherosclerosis (Vascular disorders) | 0 (0) | 1 (1) | NA | NA
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optilume™ BPH Catheter Treatment in Men With Symptomatic BPH System (N=98) | Sham BPH Catheter Treatment in Men With Symptomatic BPH. (N=48) | Crossover Cohort (N=25) | Pharmacokinetic(PK) (N=14)
Hemorrhoids (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 17 (17) | 6 (6) | 2 (2) | 0 (0)
Elevated Prostate Specific Antigen (PSA) (Investigations) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 9 (9) | 1 (1) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 14 (14) | 2 (2) | 0 (0) | 1 (1)
Lower Urinary Tract (Renal and urinary disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Post Procedural Hematuria (Renal and urinary disorders) | 30 (30) | 0 (0) | 6 (6) | 1 (1)
Stress Urinary Incontinence (Renal and urinary disorders) | 7 (7) | 0 (0) | 1 (1) | 1 (1)
Urinary Incontinence (Urge/Mixed) (Renal and urinary disorders) | 8 (8) | 1 (1) | 4 (4) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04131907/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT04131907/SAP_001.pdf